CLINICAL TRIAL: NCT01934439
Title: AMES Rehabilitation of the Proximal Arm in Severely Impaired Stroke Patients
Brief Title: AMES Treatment of the Proximal Arm in Chronic Stroke
Acronym: AMES
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Loss of funding; could not complete building the testing device.
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Paul J. Cordo, Sub-Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00009262; OCF9009196 (Other: Oregon Community Foundation)
Record Dates: First submitted 2013-08-26; First posted 2013-09-04 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: Stroke; Rehabilitation; Dyssynergia; Robotics; AMES; Cerebrovascular Accident
MeSH Terms: conditions — Stroke; Ataxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PAAD (Proximal Arm AMES Device)Treatments (Experimental): The PAAD flexes and extends the elbow, and it abducts and adducts the shoulder, where "abduction" is away from the side of the body, and "adduction" is towards it. Elbow extension occurs simultaneously with shoulder abduction, and elbow flexion occurs simultaneously with shoulder adduction. At the same time as the movements, vibrators are utilized to activate muscle spindle Ia receptors in the muscles of the arm to exaggerate the perception of movement.
  Interventions: Device: 30 PAAD treatments

INTERVENTIONS:
Device: 30 PAAD treatments — Subjects will don a shirt with pockets at the elbow and shoulder in each of which a muscle vibrator is located. The subject will then place the affected arm in the PAAD. The PAAD will range the affected arm, at the shoulder in the adduction-abduction direction, and at the elbow in the flexion-extension direction. The subject will assist volitionally this motion, and visual feedback of the level of their assistive torque will be provided along with a target torque level. The muscle vibrators will alternate from one side of each of the 2 joints to the other as the motion reverses, vibration always being applied to the lengthening muscles. This treatment will last 30 min in each session.

SUMMARY:
Subjects will receive 30 treatments with AMES, to the proximal arm which has been affected by a chronic stroke.

DETAILED DESCRIPTION:
This study seeks to determine whether 30 treatments with AMES, to the proximal affected arm of subjects with chronic stroke, will improve subjects' proximal arm active range-of-motion. We hypothesize that the combination of assisted movement, torque biofeedback, and muscle vibration will reduce impairment (i.e., increase strength and range-of-motion; decrease inappropriate patterns of muscle contraction) and, thereby, lead to more accurate reaching with the proximal arm.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or Hemorrhagic stroke affecting the right arm
* One year or longer since stroke
* Severe impairment of right arm with a baseline upper extremity Fugl-Meyer score between 8-24
* Right elbow and shoulder spasticity (Ashworth score ≤3)
* Right shoulder abduction-elbow flexion dyssynergia

Exclusion Criteria:

* Exercise intolerance
* Co-morbidities limiting arm movement (e.g. shoulder subluxation)
* Chronic pain
* Cognitive dysfunction preventing compliance with instructions
* Participation in other ongoing research studies
* Plans to initiate or discontinue any physical/occupational therapy during the period of enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment - Upper Extremity | Baseline and change from baseline at 0 and 3 months post completion

SECONDARY OUTCOMES:
Ashworth Spasticity Scale | Baseline and change from baseline at 0 and 3 months post completion
Modified Wolf Motor Test | Baseline and change from baseline at 0 and 3 months post completion

OTHER OUTCOMES:
Box and Block Test | Baseline and change from baseline at 0 and 3 months post completion
Upper extremity strength of the shoulder and elbow joints | Baseline, after each of 30 treatments, 3 months post completion of all treatments
  The PAAD measures the strength at the elbow and shoulder by recording the torque applied by the subject to the device with the elbow and shoulder during maximal efforts.
Reaching Test | Baseline and change from baseline at 0 and 3 months post completion
  In the Reaching Test, a video system will test each participant's pointing accuracy and smoothness of transportation of the arm to reach specific targets.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Oken, MD, Principal Investigator — Oregon Health and Science University; Paul J Cordo, Ph.D, Study Director — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University West Campus, Beaverton, Oregon, United States

REFERENCES:
- [Background] Cordo P, Lutsep H, Cordo L, Wright WG, Cacciatore T, Skoss R. Assisted movement with enhanced sensation (AMES): coupling motor and sensory to remediate motor deficits in chronic stroke patients. Neurorehabil Neural Repair. 2009 Jan;23(1):67-77. doi: 10.1177/1545968308317437. Epub 2008 Jul 21. PMID 18645190